CLINICAL TRIAL: NCT02924558
Title: Metabolic Effects of Replacing Dietary Refined Carbohydrate With a Combination of Egg Protein and Unsaturated Fats in Men and Women With Elevated Triglycerides
Brief Title: Metabolic Effects of Egg Protein and Unsaturated Fat Intakes in Subjects With Hypertriglyceridemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: American Egg Board (Other); Egg Nutrition Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MC-1412
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Hypertriglyceridemia
Keywords: Egg; Protein; Unsaturated fatty acids; Triglycerides; Insulin sensitivity; Lipid triad
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance | interventions — Egg Proteins; Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egg protein/unsaturated fatty acid (Experimental): 8% higher protein energy (from egg protein) and 8% higher fat energy (from unsaturated fatty acids); approximately 42/23/35% kcal from carbohydrate/protein/fat, respectively
  Interventions: Other: Egg protein/unsaturated fatty acid
- Control (Placebo Comparator): 16% higher carbohydrate energy; approximately 58/15/27% kcal from carbohydrate/protein/fat, respectively
  Interventions: Other: Control

INTERVENTIONS:
Other: Egg protein/unsaturated fatty acid — Study test foods (yogurt, muffins, waffles, and cookies) containing 8% higher protein energy (egg protein) and 8% higher fat energy (unsaturated fatty acids) than Control
  Arms: Egg protein/unsaturated fatty acid
Other: Control — Study test foods (yogurt, muffins, waffles, and cookies) containing 16% higher carbohydrate energy than Egg protein/unsaturated fatty acid
  Arms: Control

SUMMARY:
The goal of this study is to evaluate the effects of replacing some refined starches and added sugars with a combination of egg protein and unsaturated fatty acids on markers of cardiometabolic health in men and women with hypertriglyceridemia.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effects of a combination of egg protein and unsaturated fatty acids acting as substitutes for ~16% of energy from refined carbohydrate on the metabolic profile of men and women with elevated triglycerides. This is a randomized, controlled feeding, crossover trial that includes two screening/baseline visits, two 3-week treatment conditions, and a 2-week washout phase. Subjects consume a standardized background diet (7-day rotating menu) that incorporates at least 3 servings/day of study test foods, providing 40-60% of subjects' daily energy needs. Study test foods consist of yogurt, muffins, waffles, and cookies. The test foods account for 8% higher protein energy (from egg protein) and 8% higher fat energy (from unsaturated fatty acids) in the Active Condition compared to the Control Condition. In the Control Condition, the study foods account for 16% higher carbohydrate energy. The overall macronutrient composition of each condition is as follows: Active Condition, approximately 42/23/35% kcal from carbohydrate/protein/fat, respectively, and Control Condition, approximately 58/15/27% kcal from carbohydrate/protein/fat, respectively. Blood samples will be collected at baseline and end of treatment for measurement of metabolic parameters, and a liquid meal tolerance test (LMTT) will be conducted at baseline and the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Fasting TG level 150-499 mg/dL
* Body mass index (BMI) 25.0-39.9 kg/m2
* Score of 7-10 on Vein Access Scale
* Normally active and judged to be in general good health on basis of medical history and routine laboratory tests

Exclusion Criteria:

* Fasting blood glucose ≥126 mg/dL or known type 1 or type 2 diabetes mellitus
* Atherosclerotic cardiovascular disease
* Recent history or current significant renal, pulmonary, hepatic, biliary, or gastrointestinal disease
* Abnormal lab test results of clinical significance (e.g., creatinine ≥1.5 mg/dL and aspartate or alanine transaminase ≥1.5 times upper limit of normal)
* History of cancer in previous 2 years
* Uncontrolled hypertension
* Recent unstable use of anti-hypertensive medication, thyroid hormone replacements, and/or medications known to substantially influence carbohydrate metabolism
* Recent use of certain blood pressure medications (e.g., beta-adrenergic blockers and/or high-dose thiazide diuretics)
* Recent use of lipid-altering drugs (e.g., statins, bile acid sequestrants, cholesterol absorption inhibitors, or fibrates)
* Recent use of diabetes medication (e.g., alpha-glucosidase inhibitors, biguanides and biguanide combinations, bile acid sequestrants, thiazolidinediones, dipeptidyl peptidase-4 inhibitors, meglitinides, and sulfonylureas and combination sulfonylureas)
* Recent use of lipid-altering foods, herbs, or dietary supplements (e.g., niacin, sterol/stanol products, dietary fiber supplements, red rice yeast supplements)
* Recent unstable use of herbs and dietary supplements that may influence carbohdyrate metabolism
* Extreme dietary habits, dietary restrictions, or significant food allergies
* Required energy intake <2200 kcal/day or >3400 kcal/day
* Recent change in body weight of ±4.5 kg
* Recent use of weight loss drugs or programs
* Active infection or on antibiotic therapy
* Current or recent history of drug or alcohol abuse
* Pregnant, planning to be pregnant, or lactating females or women of childbearing potential unwilling to commit to use of a medically approved form of contraception

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Matsuda composite index of insulin sensitivity (MISI) | 3 weeks
  Difference between treatments in percent change from baseline to end of treatment MISI calculated from glucose and insulin responses to the LMTT at Visit 2, Day 0 (baseline); Visit 6, Day 21 (end of treatment period I); and Visit 11, Day 21 (end of treatment period II)

SECONDARY OUTCOMES:
Lipoprotein lipids | 3 weeks
  Difference between treatments in percent change from baseline to end of treatment fasting triglycerides (TG), total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), non-high-density lipoprotein cholesterol (non-HDL-C), low-density lipoprotein cholesterol (LDL-C), and TC/HDL-C ratio based on the average of values collected at Visits 1 and 2, Days -7 and 0 (baseline); Visits 5 and 6, Days 19 and 21 (end of treatment period I); and Visits 10 and 11, Days 19 and 21 (end of treatment period II)
Lipoprotein particle concentrations | 3 weeks
  Difference between treatments in change from baseline to end of treatment lipoprotein particle subclass concentrations and sizes, as well as cholesterol carried by major lipoproteins and subfractions analyzed using an ion mobility assay at Visit 2, Day 0 (baseline); Visit 6, Day 21 (end of treatment period I); and Visit 11, Day 21 (end of treatment of period II)
Apolipoprotein (Apo) B | 3 weeks
  Difference between treatments in percent change from baseline to end of treatment apo B at Visit 2, Day 0 (baseline); Visit 6, Day 21 (end of treatment period I); and Visit 11, Day 21 (end of treatment period II)
Homeostasis model assessment of insulin sensitivity (HOMA2-%S) | 3 weeks
  Difference between treatments in change from baseline to end of treatment HOMA2-%S calculated from fasting values of insulin and glucose at Visit 2, Day 0 (baseline); Visit 6, Day 21 (end of treatment period I); and Visit 11, Day 21 (end of treatment period II)
LMTT disposition index | 3 weeks
  Difference between treatments in the percent change from baseline to end of treatment LMTT disposition index calculated from insulin and glucose responses during the LMTT at Visit 2, Day 0 (baseline); Visit 6, Day 21 (end of treatment period I); and Visit 11, Day 21 (end of treatment period II)
Homeostasis model assessment of pancreatic beta-cell function (HOMA2%B) | 3 weeks
  Difference between treatments in change from baseline to end of treatment HOMA2%B calculated from fasting insulin and glucose values at Visit 2, Day 0 (baseline); Visit 6, Day 21 (end of treatment period I); and Visit 11, Day 21 (end of treatment period II)
Blood pressure | 3 weeks
  Difference between treatments in change from baseline to end of treatment in systolic and diastolic blood pressures based on the average of values collected at Visits 1and 2, Days -7 and 0 (baseline); Visits 5 and 6, Days 19 and 21 (end of treatment period I); and Visits 10 and 11, Days 19 and 21 (end of treatment period II)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Principal Investigator — Midwest Center for Metabolic and Cardiovascular Research

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maki KC, Palacios OM, Lindner E, Nieman KM, Bell M, Sorce J. Replacement of Refined Starches and Added Sugars with Egg Protein and Unsaturated Fats Increases Insulin Sensitivity and Lowers Triglycerides in Overweight or Obese Adults with Elevated Triglycerides. J Nutr. 2017 Jul;147(7):1267-1274. doi: 10.3945/jn.117.248641. Epub 2017 May 17. PMID 28515160